CLINICAL TRIAL: NCT02672332
Title: A Phase 3 Multi-Center, Randomized, Double-Blinded, Vehicle-Controlled, Parallel Group Study Comparing the Efficacy, Tolerability and Safety of SB204 and Vehicle Gel Once Daily in the Treatment of Acne Vulgaris
Brief Title: P3 Study in Acne Comparing Once Daily SB204 and Vehicle
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI-AC301
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — berdazimer sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SB204 4% (Experimental): SB204 4% topically once daily
  Interventions: Drug: SB204 4%
- Vehicle Gel (Placebo Comparator): Vehicle Gel topically once daily
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: SB204 4% — Once daily
  Other Names: NVN1000
  Arms: SB204 4%
Drug: Vehicle Gel — Placebo comparator
  Other Names: Placebo
  Arms: Vehicle Gel

SUMMARY:
This is a 12 week, multi-center, double-blinded, randomized, vehicle-controlled, parallel group, study to be conducted in approximately 1300 subjects with acne vulgaris in the US.

DETAILED DESCRIPTION:
This is a double-blind, placebo controlled study in subjects with moderate to severe acne. Subjects who satisfy the entry criteria will be randomized to SB204 4% QD or Vehicle Gel QD in a 1:1 ratio. Efficacy assessments will include Investigator Global Assessments (IGA) and inflammatory and non-inflammatory lesion counts. Subjects will return for post-Baseline evaluation at Weeks 2, 4, 8, and 12/Early Termination (ET).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe acne
* Minimum of 25 and no more than 70 non-inflammatory lesions (open and closed comedones) on the face
* Minimum of 20 and no more than 40 inflammatory lesions (papules and pustules)

Exclusion Criteria:

* Women of child-bearing potential who are pregnant, nursing, considering becoming pregnant
* Any dermatologic condition that could interfere with clinical evaluations including severe, recalcitrant cystic acne

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1307 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Rico, MD, Study Chair — Novan, Inc.
Locations (55):
- United States (55):
  - CIL #146, Anaheim, California
  - CIL #118, Encinitas, California
  - CIL #186, Fresno, California
  - CIL #210, Fresno, California
  - CIL #209, Oceanside, California
  - CIL #161, San Diego, California
  - CIL #113, San Diego, California
  - CIL #199, Santa Rosa, California
  - CIL #103, Boca Raton, Florida
  - CIL #173, Hialeah, Florida
  - CIL #212, Homestead, Florida
  - CIL #222, Lauderdale Lakes, Florida
  - CIL #157, Miami, Florida
  - CIL #177, North Miami Beach, Florida
  - CIL #150, Orlando, Florida
  - CIL #172, Orlando, Florida
  - CIL #203, Ormond Beach, Florida
  - CIL #211, South Miami, Florida
  - CIL #229, Tampa, Florida
  - CIL #153, Wellington, Florida
  - Cil # 179, Chicago, Illinois
  - CIL #215, Wichita, Kansas
  - CIL #117, Louisville, Kentucky
  - CIL #180, New Orleans, Louisiana
  - CIL #205, Glenn Dale, Maryland
  - CIL #230, Quincy, Massachusetts
  - CIL #112, Detroit, Michigan
  - CIL #149, Troy, Michigan
  - CIL #225, Saint Joseph, Missouri
  - CIL #187, St Louis, Missouri
  - CIL #140, Omaha, Nebraska
  - CIL #182, Las Vegas, Nevada
  - CIL #201, Berlin, New Jersey
  - CIL #141, Montclair, New Jersey
  - CIL #156, Albuquerque, New Mexico
  - CIL #107, New York, New York
  - CIL #108, Rochester, New York
  - CIL #104, Stony Brook, New York
  - CIL #193, High Point, North Carolina
  - CIL #166, Winston-Salem, North Carolina
  - CIL #226, Cincinnati, Ohio
  - CIL #200, Portland, Oregon
  - CIL #236, Charleston, South Carolina
  - CIL #217, Chattanooga, Tennessee
  - CIL #198, Arlington, Texas
  - CIL #154, Beaumont, Texas
  - CIL #162, Carrollton, Texas
  - CIL #188, Houston, Texas
  - CIL #151, Plano, Texas
  - CIL #168, Plano, Texas
  - CIL #224, San Antonio, Texas
  - CIL #171, San Antonio, Texas
  - CIL #164, Sugar Land, Texas
  - CIL #106, Salt Lake City, Utah
  - CIL #114, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1300 participants were planned to be recruited from dermatologists and other (e. g. family physicians, research clinics). A total of 1307 participants were randomized. Enrollment began on 22Feb2016 and the last subject completed on 21Dec2016. There were 1306 participants in the intent to treat (ITT) and safety populations.
Groups:
- Vehicle Gel: Vehicle Gel (placebo comparator) topically once daily
Period: Overall Study
Arm/Group | SB204 4% | Vehicle Gel
Started | 653 | 654
Completed | 571 | 577
Not Completed | 82 | 77

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population: all study subjects who were randomized and dispensed study medication, and were grouped by the treatment the subject was assigned to at the time of randomization. There were 653 subjects randomized to SB204, but one subject was excluded from the ITT due to not meeting inclusion/exclusion criteria, thereby reducing the Baseline ITT population for SB204 to 652. All efficacy analyses were performed on the ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | SB204 4% | Vehicle Gel | Total
Number analyzed (Participants) | 652 | 654 | 1306
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.1 (8.25) | 21.3 (8.38) | 21.2 (8.32)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject was excluded from the ITT after randomization, prior to receiving study medication due to not meeting inclusion/exclusion criteria.
  Participants
    Female | 400 | 406 | 806
    Male | 252 | 248 | 500
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One subject was excluded from the ITT after randomization, prior to receiving study medication due to not meeting inclusion/exclusion criteria.
  Participants
    American Indian or Alaska Native | 3 | 2 | 5
    Asian | 28 | 26 | 54
    Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
    Black or African American | 143 | 148 | 291
    White | 456 | 455 | 911
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 20 | 21 | 41
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 652 | 654 | 1306
Baseline Investigator Global Assessment [Count of Participants; unit: Participants] — Population: Statistical analyses were not reported for the overall study population; they were only reported for the individual treatment groups.
  Participants
    0--clear: number analyzed (Participants) | 651 | 653 | 1304
    0--clear | 0 | 0 | 0
    1--almost clear: number analyzed (Participants) | 651 | 653 | 1304
    1--almost clear | 0 | 0 | 0
    2--mild: number analyzed (Participants) | 651 | 653 | 1304
    2--mild | 0 | 0 | 0
    3--moderate: number analyzed (Participants) | 651 | 653 | 1304
    3--moderate | 557 | 575 | 1132
    4--severe: number analyzed (Participants) | 651 | 653 | 1304
    4--severe | 94 | 78 | 172

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Inflammatory Lesion Counts
Description: The absolute change from Baseline in inflammatory lesion counts was to be assessed on the face only (forehead, right and left cheeks, chin, and nose). Inflammatory lesions included papules, pustules, nodules, and cysts.
Time Frame: Baseline and Week 12
Population: Intent To Treat population (ITT)
Measure: Mean (Standard Deviation); unit: inflammatory acne lesions
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 651 | 653
inflammatory acne lesions | -12.4 (10.30) | -11.3 (10.46)

2. Primary Outcome: Absolute Change From Baseline in Non-inflammatory Lesion Counts
Description: The absolute change from Baseline in non-inflammatory lesion counts was to be assessed on the face only (forehead, right and left cheeks, chin, and nose). Non-inflammatory lesions included open comedones (blackheads) and closed comedones (whiteheads).
Time Frame: Baseline and Week 12
Population: Intent to Treat population (ITT)
Measure: Mean (Standard Deviation); unit: non-inflammatory acne lesions
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 651 | 653
non-inflammatory acne lesions | -16.0 (16.36) | -13.5 (16.97)

3. Primary Outcome: Proportion of Subjects With Investigator Global Assessment (IGA) Success at Week 12
Description: Proportion of subjects with Investigator Global Assessment (IGA) Success at Week 12 is defined as an IGA score of 0 or 1 (Clear/Almost Clear) and at least a 2 grade improvement from Baseline. The IGA scale is as follows:
  Grade Description 0 Clear: Clear skin with no inflammatory or non-inflammatory lesions.
  1. Almost clear: Rare non-inflammatory lesions with rare papules (papules may be resolving and hyperpigmented, though not pink-red).
  2. Mild: Some non-inflammatory lesions with no more than a few inflammatory lesions.
  3. Moderate: Up to many non-inflammatory lesions and may have some inflammatory lesions, but no more than one nodulocystic lesion.
  4. Severe: Up to many non-inflammatory and inflammatory lesions, but no more than a few nodulocystic lesions
Time Frame: Baseline and Week 12
Population: ITT population; subjects who had a Week 12 (study completion) visit.
Measure: Count of Participants; unit: Participants
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 599 | 592
Participants | 83 | 84

4. Secondary Outcome: Percent Change in Inflammatory Lesion Count
Description: The percent change from baseline in inflammatory lesion count
Time Frame: Baseline and Week 12
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 651 | 653
Percentage change from baseline | -45.9 (36.65) | -43.1 (38.68)

5. Secondary Outcome: Percent Change in Non-inflammatory Lesion Count
Description: The percent change from baseline in non-inflammatory lesion count
Time Frame: Baseline and Week 12
Population: ITT population
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 651 | 653
Percentage change from baseline | -39.6 (35.84) | -34.6 (41.82)

6. Secondary Outcome: Time to Reduction in Inflammatory Lesion Counts
Description: Median time to a 35% reduction in inflammatory lesion count (Kaplan-Meier)
Time Frame: Week 12
Population: ITT population; overall number of participants analyzed = the # of participants who achieved at least a 35% reduction in their inflammatory lesion counts.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 506 | 494
Days | 31.0 [30.0 to 37.0] | 31.0 [29.0 to 55.0]

7. Secondary Outcome: Time to Improvement in IGA
Description: Median time to a 2 or more grade improvement in IGA (Kaplan-Meier analysis).
Time Frame: Week 12
Population: ITT population. Overall number of participants analyzed = number of participants who achieved a 2 or more grade improvement in their IGA score. This was a Kaplan-Meier analysis; for both the SB204 4% and Vehicle Gel treatment groups, the median was not estimable due to < 50% of subjects achieving a 2 or more grade improvement in their IGA score.
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | SB204 4% | Vehicle Gel
Number analyzed (Participants) | 133 | 120
Days
  25% Quartile | 87.0 [86.0 to 90.0] | 87.0 [86.0 to NA] — The upper bounds of the CI is not available because not enough subjects achieved a 2 or more grade improvement in their IGA score prior to their last visit.
  50% Quartile | NA [NA to NA] — The median was not estimable due to < 50% of subjects achieving a 2 or more grade improvement in their IGA score. | NA [NA to NA] — The median was not estimable due to < 50% of subjects achieving a 2 or more grade improvement in their IGA score.
  75% Quartile | NA [NA to NA] — The median was not estimable due to < 50% of subjects achieving a 2 or more grade improvement in their IGA score. | NA [NA to NA] — The median was not estimable due to < 50% of subjects achieving a 2 or more grade improvement in their IGA score.

ADVERSE EVENTS:
Time Frame: Adverse events were collected after the subject signed the informed consent and completed any study assessment until the end of the final study visit, approximately 12 weeks for most subjects.
Description: Adverse events were collected for all subjects who were randomized and received at least one dose of study medication. Two subjects who were randomized to the Vehicle group received SB204 and per the definition of the Safety Population in the Statistical Analysis Plan, these subjects were analyzed in the SB204 group. Therefore, 654 subjects were in the SB204 group and 652 subjects were in the Vehicle group for analyses of all cause mortality, adverse events and serious adverse events.
Arm/Group | SB204 4% | Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 0/654 | 1/652
Serious Adverse Events (participants affected / at risk) | 0/654 | 4/652
Other Adverse Events (participants affected / at risk) | 66/654 | 10/652
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB204 4% (N=654) | Vehicle Gel (N=652)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) — Subject was a 66 year old male; died of natural causes (unknown) and the event was considered to be not related to treatment
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Bulimia nervosa (Psychiatric disorders) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SB204 4% (N=654) | Vehicle Gel (N=652)
Application site pain (General disorders) | 21 | 3
Application site pruritus (General disorders) | 16 | 3
Nasopharyngitis (Infections and infestations) | 11 | 10
Application site erythema (General disorders) | 11 | 1
Application site dryness (General disorders) | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-01-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT02672332/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT02672332/SAP_001.pdf